CLINICAL TRIAL: NCT07383519
Title: Dahua Hospital, Xuhui District, Shanghai
Brief Title: Application of Photon Therapy Instrument Combined With Ultrasonic Debridement in Senile Third and Fourth Stage Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dahua Hospital, Xuhui District, Shanghai (Other Government)
Responsible Party: Principal Investigator, Jie Zeng, Dahua Hospital, Xuhui District, Shanghai, Dahua Hospital, Xuhui District, Shanghai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20220603
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2023-05

CONDITIONS: Photon Therapy; Ultrasonic Debridement; Combination Therapy; Geriatric Patients; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photon Therapy Combined with Ultrasonic Debridement Group (Other): Participants in this arm received the combined intervention of ultrasonic debridement followed by photon therapy in addition to standard moist wound care and systemic management. Ultrasonic debridement was performed using a handheld device held at a 45-degree angle approximately 0.5 cm from the wound surface to selectively remove necrotic tissue. Subsequently, photon therapy was administered with the light source positioned 10 cm from the wound for 15 minutes per session, using blue light (for infected wounds) followed by red light as indicated. This combined physical therapy regimen aimed to enhance wound bed preparation, reduce bacterial load, promote tissue repair, and accelerate healing in elderly patients with stage 3 or 4 pressure injuries.
  Interventions: Other: Photon Therapy Combined with Ultrasonic Debridement Group
- Standard Wound Care Grou (Other): Participants in this arm received standard moist wound care guided by the TIME principle (Tissue management, Infection/inflammation control, Moisture balance, and Edge advancement) and systemic interventions. Wounds were cleansed with 0.9% normal saline, and appropriate dressings were selected based on wound stage and exudate level. Dressing change frequency was determined according to clinical need. Systemic factors affecting wound healing were addressed, and comprehensive health education was provided, including guidance on repositioning, nutrition, and home care. This arm served as the control to evaluate the added benefit of the combined physical therapy intervention.
  Interventions: Other: Standard Wound Care Group

INTERVENTIONS:
Other: Photon Therapy Combined with Ultrasonic Debridement Group — Participants in this arm received the combined intervention of ultrasonic debridement followed by photon therapy in addition to standard moist wound care and systemic management. Ultrasonic debridement was performed using a handheld device held at a 45-degree angle approximately 0.5 cm from the wound surface to selectively remove necrotic tissue. Subsequently, photon therapy was administered with the light source positioned 10 cm from the wound for 15 minutes per session, using blue light (for infected wounds) followed by red light as indicated. This combined physical therapy regimen aimed to enhance wound bed preparation, reduce bacterial load, promote tissue repair, and accelerate healing in elderly patients with stage 3 or 4 pressure injuries.
  Arms: Photon Therapy Combined with Ultrasonic Debridement Group
Other: Standard Wound Care Group — Participants in this arm received standard moist wound care guided by the TIME principle (Tissue management, Infection/inflammation control, Moisture balance, and Edge advancement) and systemic interventions. Wounds were cleansed with 0.9% normal saline, and appropriate dressings were selected based on wound stage and exudate level. Dressing change frequency was determined according to clinical need. Systemic factors affecting wound healing were addressed, and comprehensive health education was provided, including guidance on repositioning, nutrition, and home care. This arm served as the control to evaluate the added benefit of the combined physical therapy intervention.
  Arms: Standard Wound Care Grou

SUMMARY:
These findings support the integrated use of ultrasonic debridement and photon therapy as a beneficial treatment strategy for advanced pressure injuries in elderly patients, demonstrating its value in improving both clinical results and overall patient well-being.

DETAILED DESCRIPTION:
This study assessed the clinical effectiveness of combining ultrasonic debridement with photon therapy for treating stage 3 and 4 pressure injuries in elderly patients, with particular attention to wound healing, pain reduction, and quality of life outcomes. We enrolled 118 elderly patients with pressure injuries from Shanghai Dahua Hospital between May 1, 2023, and November 30, 2024, using stratified random sampling. Participants were first grouped by injury stage (3 or 4) and then randomly assigned to either control or experimental groups. Control patients received standard moist wound care alongside systemic interventions, whereas the experimental group received the same standard care plus combined ultrasonic debridement and photon therapy. We compared outcomes including wound healing progress, treatment expenses, and pain scores recorded during dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* age 55 years or older
* a patient who is fully conscious (i.e., no disturbance of consciousness such as drowsiness, lethargy, or delirium; able to accurately answer questions about time, place, and person orientation; and capable of clear communication to express needs or understand study-related instructions)
* patients with pressure injury were diagnosed with stage 3 or 4 pressure injury in accordance with the staging criteria of pressure injury published by the National Pressure Injury Advisory Panel (NPUAP).

Exclusion Criteria:

* poor blood glucose control (HbA1c > 7.0%)
* patients allergic to red-and-blue light
* mental abnormalities who cannot cooperate with treatment
* patients with advanced malignancies, terminal patients, patients with cachexia, and patients with severe obesity
* severe complications: severe malnutrition, severe diseases of the lungs, liver, kidneys, and cardiovascular system
* patients undergoing other treatments, such as Chinese medicine treatment, negative pressure aspiration therapy, platelet-rich therapy
* who were unwilling to participate in the study. All participants signed a written informed consent form before the study began.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Complete Wound Healing | Assessed at 6 months post-randomization.
  The primary outcome is the proportion of participants achieving complete wound healing, defined as a Pressure Ulcer Scale for Healing (PUSH) score of 0. The PUSH tool assesses wound area, exudate amount, and tissue type, with a total score range of 0-17.

SECONDARY OUTCOMES:
Change in Pain Intensity During Dressing Changes | Baseline and 1 month post-intervention.
  Mean change in pain scores measured using the Numeric Pain Intensity Scale (NPIS, 0-10) during dressing changes. Scores are recorded at enrollment and 1 month post-intervention.
Total Direct Medical Cost of Treatment | From randomization to 6 months post-intervention.
  The total direct medical costs (in CNY) associated with pressure injury treatment per participant, including materials, procedures, and related care, calculated over the 6-month study period.
Change in Wound Severity as Measured by the Pressure Ulcer Scale for Healing (PUSH) Score | Baseline, 1 month, 3 months, and 6 months post-intervention.
  Mean change in PUSH scores from baseline to 1, 3, and 6 months post-intervention. A reduction in score indicates wound improvement.

OTHER OUTCOMES:
Complete Healing Rate Stratified by Pressure Injury Stage | 3 months and 6 months post-intervention.
  The proportion of participants achieving complete wound healing (PUSH = 0) separately for stage 3 and stage 4 pressure injuries at 3 and 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Dahua Hospital, Xuhui District, Shanghai, Shanghai, Shanghai Municipality, China